CLINICAL TRIAL: NCT05090488
Title: The Integration of Health Coaching and Diabetes Education in Type 2 Diabetes Mellitus Patients at Jakarta Primary Health Care: Role on Metabolic Control, Diabetes Complications, Inflammatory Marker, Behavior Changes, and Quality of Life
Brief Title: Integration of Health Coaching and Diabetes Education in Type 2 Diabetes Mellitus Management at Primary Health Care
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Indonesia University (Other)
Collaborators: Provincial Health Services Authority British Columbia (Other)
Responsible Party: Principal Investigator, Em Yunir, DR. dr. Em Yunir, SpPD, KEMD, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Health Coaching Jakarta
Record Dates: First submitted 2021-02-11; First posted 2021-10-22 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Type2 Diabetes; Diabetes Mellitus, Type 2; Endocrine System Diseases; Nutritional and Metabolic Diseases; Glucose Metabolism Disorders (Including Diabetes Mellitus); Diabetes Mellitus
Keywords: Type 2 Diabetes Mellitus; Diabetes Education; Health Coaching
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Endocrine System Diseases; Nutritional and Metabolic Diseases; Glucose Metabolism Disorders; Diabetes Mellitus | interventions — Population Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Received Personal Health Coaching and Diabetes Education in Group (Experimental): Health coaching was given as face to face with a trained coach from primary health care. Diabetes education in group, with trained educator team from primary health care
  Interventions: Behavioral: Personal Health Coaching and Diabetes Education in Group
- Received Diabetes Education in Group (Active Comparator): Diabetes education in group, with trained educator team from primary health care
  Interventions: Behavioral: Personal Health Coaching and Diabetes Education in Group

INTERVENTIONS:
Behavioral: Personal Health Coaching and Diabetes Education in Group — Health coaching was given as face to face with a trained coach from primary health care. Diabetes education in group, with trained educator team from primary health care

SUMMARY:
Type 2 Diabetes Mellitus is a chronic disease with increasing incidence globally. It needs a comprehensive and continuous management approach that includes five pillars: education, nutritional management, physical activity, pharmacological treatment, and monitoring. To achieve good glycemic control, prevention of complications, and good quality of life as diabetes management goals, patients' capability to properly navigate diabetes management is a key. One evidence-based model to empower patients' self-management abilities is diabetes education and health coaching. Diabetes management at primary health care needs special concern since they play an important role in initial and continuing care for diabetes patients in the community. Therefore, the implementation of diabetes education and health coaching in primary health care is expected to improve the self-management abilities of people with diabetes

DETAILED DESCRIPTION:
A randomized control trial, pre and post study involving 180 subjects randomized into 2 arms:

* Control : received education in group
* Intervention : received education group + personal health coaching Education group divided into 6 session, which for each session consist of 2 different topics and lasts for 60 minutes.

Health coaching was given by a coach, a healthcare professional who undergo training to become a coach. Health coaching delivered as face to face between subjects and coach.

Laboratory examination, anthropometric measurement, echocardiography, electrocardiography, Heart Rate Variability measurement, diabetic eye screening, and questionnaire collected at baseline, 3 and 6 months after intervention

ELIGIBILITY:
Inclusion Criteria:

* Type 2 Diabetes Mellitus
* >= 18 years old
* Willing to follow the research by signing an informed consent

Exclusion Criteria:

* Patients with cognitive disease (such as dementia)
* Patients with hearing or sight problem
* Unable to live independently on daily basis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-12-14 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Change from baseline HbA1C at 3 months and 6 months | Baseline, 3 and 6 months after intervention
  HbA1C is indicator of glycemic control

SECONDARY OUTCOMES:
Change from baseline fasting plasma glucose at 3 and 6 months | Baseline, 3 and 6 months after intervention
  Blood glucose monitoring
Change from baseline serum lipid at 3 and 6 months | Baseline, 3 and 6 months after intervention
  Lipid profile measurement includes total cholesterol, LDL-cholesterol, HDL-cholesterol, and triglycerides
Change from baseline inflammatory marker at 3 and 6 months | Baseline, 3 and 6 months after intervention
  Inflammatory marker used is hs-CRP (C-reactive protein)
Change from baseline body mass index | Baseline, 3 and 6 months after intervention
  Body mass index described by kg/m2
Change from baseline waist circumference | Baseline, 3 and 6 months after intervention
  Waist circumference measured by cm
Change from baseline body fat | Baseline, 3 and 6 months after intervention
  Body fat measured by body impedance analysis
Change from baseline left ventricular mass index | Baseline, 6 months after intervention
  Left ventricular mass index measured using standard formula and corrected by body surface area
Change from baseline left ventricular systolic function | Baseline, 6 months after intervention
  Left ventricular systolic funciton was calculated from ejection fraction and global longitudinal strain (measured by echocardiography)
Change from baseline left atrial volume | Baseline, 6 months after intervention
  Left atrial volume was measured through biplane area calculation in echocardiography procedure
Change from baseline right ventricular systolic function | Baseline, 6 months after intervention
  Right ventricular systolic function was evaluated using TAPSE
change from baseline left ventricular diastolic function | Baseline, 6 months after intervention
  LV diastolic function was evaluated according to algorithm recommended by American Society of Echochardiography in 2016
Change from baseline electrocardiography pattern | Baseline and 6 months after intervention
  Electrocardiography pattern was used to analyze cardiac rythm
Change from baseline heart rate variability | Baseline and 6 months after intervention
  Heart rate variability was measured using ECG Holter examination
Baseline visual acuity | Baseline
  Visual acuity was measured by Peek acuity chart application using WHO classification
Baseline lens haziness | Baseline
  Lens haziness was evaluated using shadow test
Baseline retina examination | Baseline
  Retina was examined using funduscopic photography
Baseline intraocular pressure | Baseline
  Intraocular pressure was measured by cup-to-disc ratio using funduscopic photograpy
Change from baseline peripheral sensory neuropathy | Baseline, 3 and 6 months after intervention
  Peripheral sensory neuropathy was measured using combination of subjective manifestation, 10 g Simme Weinstein monofilament and 128 Hz tuning fork
Change from baseline peripheral autonomic neuropathy | Baseline, 3 and 6 months after intervention
  Peripheral autonomic neuropathy was seen visually by objective examination (dry, scaly skin and cracked skin)
Change from baseline peripheral motor neuropathy | Baseline, 3 and 6 months after intervention
  Peripheral motor neuropathy was seen visually by objective examination (changes in the shape of fingers, muscle atrophy, or bone protrusions)
Change from baseline peripheral arterial disease | Baseline, 3 and 6 months after intervention
  Peripheral arterial disease was diagnosed through ankle brachial index measurement
Change from baseline renal function | Baseline and 6 months after intervention
  Renal function was measured by estimated glomerular filtration rate (eGFR) using creatinine data
Change from baseline albuminuria | Baseline and 6 months after intervention
  Albuminuria was measured by albumin creatinine ratio
Change from baseline mean calorie intake | Baseline, 3 and 6 months after intervention
  Evaluation of mean calorie intake using food record data
Change from baseline global physical activity | Baseline, 3 and 6 months after intervention
  Global physical activity was evaluated by global physical activity questionnaire
Change from baseline medication adherence | Baseline, 3 and 6 months
  Medication adherence was measured by Morisky Medication Adherence Scale (MMAS)
Change from baseline quality of life | Baseline, 3 and 6 months
  Quality of life was evaluated by EuroQol five-dimensional questionnaire. This questionnaire evaluates 5 dimensions of life. Each dimension scores 1-5 (1 means no problem and 5 means extreme problems).

CONTACTS AND LOCATIONS:
Overall Officials: Em Yunir, PhD, Principal Investigator — Divisi Metabolik Endokrin IPD FKUI RSCM
Locations (1):
- University of Indonesia, Jakarta, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No